CLINICAL TRIAL: NCT00760058
Title: Visual Outcome and Visual Quality After Bilateral Implantation of the AcrySof® IQ IOL Compared to MI60® and Tecnis® IOL
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Enrollment not initiated for study.
Sponsor: Alcon Research (Industry)
Responsible Party: Robert Kitchen, Director of Scientific Affairs, Alcon Laboratories (Australia) Pty Ltd
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AUS-06-02
Record Dates: First submitted 2008-09-24; First posted 2008-09-25 (Estimated); Last update posted 2015-05-12 (Estimated); Status verified 2010-03

CONDITIONS: Cataract
Keywords: cataract, intraocular lens
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): AcrySof® IQ intraocular lens
  Interventions: Device: AcrySof® IQ IOL
- 2 (Active Comparator): Tecnis® Aspheric intraocular lens
  Interventions: Device: Tecnis® Aspheric intraocular lens
- 3 (Active Comparator): Akreos® MI60 intraocular lens
  Interventions: Device: Akreos® MI60 intraocular lens

INTERVENTIONS:
Device: AcrySof® IQ IOL — Replacement of natural crystalline lens in cataract surgery
  Arms: 1
Device: Tecnis® Aspheric intraocular lens — Replacement of natural crystalline lens in cataract surgery
  Arms: 2
Device: Akreos® MI60 intraocular lens — Replacement of natural crystalline lens in cataract surgery
  Arms: 3

SUMMARY:
The objective of the study is to compare the visual outcomes of three aspheric monofocal intraocular lenses after cataract surgery - ACRYSOF® IQ, Tecnis® and Akreos® MI60.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects, aged 50 and over.
* Subjects diagnosed with bilateral cataracts requiring cataract extraction and implantation of a posterior chamber intraocular lens.
* Subjects must be willing to undertake the additional ophthalmic tests within 3 months of the second lens implantation.
* Subjects must be assessed to be able to dilate to a minimum of 6 mm pre operatively.
* Subjects' pupil size must be ≥ 4.5 mm in mesopic conditions.

Exclusion Criteria:

* Subjects who have previously had corneal surgery.
* Subjects who have potential visual acuity which is < 6/12 due to other ocular pathology
* Subjects with corneal pathology.
* Subjects with astigmatism of greater than 1D.
* Subjects diagnosed with glaucoma.
* Subjects diagnosed with diabetes.
* Subjects who have previously participated in a clinical investigation within 30 days prior to enrolment
* Subjects with a know history of poor compliance
* Subjects with planned adjunctive surgery

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-06; Primary Completion 2010-12 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Contrast sensitivity | 3 months

SECONDARY OUTCOMES:
Visual acuity, contrast acuity, wavefront analysis, corneal spherical aberration, manifest refraction. | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Alcon Call Center, Fort Worth, Texas, United States